CLINICAL TRIAL: NCT02015364
Title: Non-operative Treatment of Acute Achilles Tendon Rupture, Early Controlled Mobilization Compared With Immobilization: A Blinded Randomized, Controlled Trial
Brief Title: Non-operative Treatment of Acute Achilles Tendon Rupture: Early Controlled Mobilization Compared With Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: DJO Incorporated (Industry); The Danish Rheumatism Association (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATR_Denmark_2014
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Achilles Tendon Rupture; Deep Vein Thrombosis
Keywords: Achilles tendon; Rupture; Rehabilitation; Dynamic rehabilitation
MeSH Terms: conditions — Venous Thrombosis; Rupture

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controlled early mobilization (Experimental): The intervention group: Must perform controlled mobilization-exercises from the beginning of week 3 to 8
  Interventions: Procedure: Controlled early mobilization
- Immobilization (No Intervention): The control group: In line with the current treatment regimen the patients must keep the boot on at all times and they are not allowed to move the ankle.

INTERVENTIONS:
Procedure: Controlled early mobilization — 1. The intervention group: Must perform controlled mobilization-exercises from the beginning of week 3 - 8.
  Arms: Controlled early mobilization

SUMMARY:
Study objectives To investigate if early controlled mobilization of the ankle in week 3 to 8 affects the functional outcome and patient reported outcome after treatment of acute Achilles tendon rupture.

Type of study

Randomized, controlled trial (RCT). 130 patients will be included.

Time schedule

Begins January 2014. Study period is 4-5 years; recruitment is expected to span 2 years

Setup At Copenhagen University Hospital Hvidovre the majority of patients with acute ATR are treated non-operatively. A cast is applied in the emergency room. After 2 weeks the bandage is changed to a removable orthosis and full weight bearing is allowed.

Patients who choose to participate in the trial will - through randomisation - be placed in one of the two groups:

1. The intervention group: Must perform controlled mobilization-exercises from the beginning of week 3.
2. The control group: In line with the current treatment regimen the patients must keep the boot on at all times and they are not allowed to move the ankle.

Treatment protocol for the two groups is similar concerning orthose, removal of wedges and weight-bearing. The only difference is that patients in the intervention group are instructed to do ankle exercise.

Post-examinations in relation to the study Follow-up is done at 8 and 16 weeks plus 6 and 12 months. The study's primary endpoint is at the 12 month mark.

Population Patients who are treated for acute Achilles tendon rupture at Copenhagen University Hospital Hvidovre. Patients who fulfil the inclusion criteria but do not wish to participate are treated according the standard regimen (non-operatively without early controlled movement of the ankle joint).

Number of patients 65 patients will be included in each group (a 130 patients in total).

DETAILED DESCRIPTION:
Study objectives To investigate if early controlled mobilization of the ankle in week 3 to 8 affects the functional outcome and patient reported outcome after treatment of acute Achilles tendon rupture.

Study Design Type of study The study is performed as a single-blinded, randomized, controlled trial (RCT). The randomisation is computer based; opaque envelopes are used. In total 130 patients will be included.

Time schedule Recruitment of patients for the study begins 1st of November 2013. The expected study period is 4-5 years; the recruitment itself is expected to span 2 years, provided that an average of 6 patients is included per month.

Method Setup At Copenhagen University Hospital Hvidovre the majority of patients with acute ATR are treated non-operatively. A cast is applied in the emergency room. After 2 weeks the bandage is changed to a removable orthosis and full weight bearing is allowed.

Patients who choose to participate in the trial will - through randomisation - be placed in one of the two groups:

1. The intervention group: Must perform controlled mobilization-exercises from the beginning of week 3.
2. The control group: In line with the current treatment regimen the patients must keep the boot on at all times and they are not allowed to move the ankle.

Treatment protocol for the two groups is similar concerning orthose, removal of wedges and weight-bearing. The only difference is that patients in the intervention group are instructed to do ankle exercise.

Compliance

The following measures will be taken to ensure compliance within the groups:

1. The intervention group: The patients will be equipped with training diaries in which they will record their training for each of the five daily training sessions.
2. The control group: The orthosis will be sealed. If the boot is removed it can be registered.

   Blinding The doctors and physical therapists who will conduct the follow-up will be blinded to the intervention. This is ensured as a Project Nurse will be in charge of the randomisation. The patients will be given a direct phone number for the Project Nurse, as he/she will be in charge of treatment related question and enquiries during the intervention period. Potential medical queries will be discussed with one of the affiliated doctors.

   Post-examinations in relation to the study Follow-up is done at 8 and 16 weeks plus 6 and 12 months. The study's primary endpoint is at the 12 month mark.

   Population Patients who are treated for acute Achilles tendon rupture at Copenhagen University Hospital Hvidovre. Patients who fulfil the inclusion criteria but do not wish to participate are treated according the standard regimen (non-operatively without early controlled movement of the ankle joint).

   Number of patients 65 patients will be included in each group (a 130 patients in total). The sample size calculation is based on a clinical relevant difference of 10 point in ATRS, a standard deviation (SD) of 16 and power of 0.90 (two sided). In a previous material, with a fully comparable population, we found a SD of 16 points at the 1 year post-examination. 54 patients is required in each group; due to the risk of drop out 65 patients will be included in each group.

   Inclusion criteria
   * Age 18-70 years.
   * The patient must be expected to be able to attend rehabilitation and post-examinations.
   * The patient must be able to speak and understand Danish.
   * The patient must be able to give informed consent. Exclusion criteria
   * Former rupture of one or both Achilles tendon(s).
   * Previous surgery on the Achilles tendon.
   * Fluoroquinolone treatment within the last 6 months.
   * Tendinosis treated with corticosteroids (tablets or injections) within the last 6 months.
   * The patient has been diagnosed with arterial insufficiency in the legs.
   * Terminal illness or severe medical illness: ASA score higher than or equal to 3.
   * The space between the rupture and the calcaneus is less than 1cm.

   Data Registration

   All relevant data is recorded in a specially designed database. The data registration will be reported to the Danish Data Protection Agency.

   Primary endpoint The primary endpoint is evaluated at 12 month.

   ATRS: Achilles tendon Total Rupture Score 25 A patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture.

   Secondary endpoints

   Heel-rise work test: Endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel-rises are counted and measured. The results are then compared to the weight of the patient and the total work is estimated. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used 25.

   Single heel-rise test: The patient stands with the foot in neutral position. It is recorded whether the patient is able to make a single heel-rise on the injured leg. The heel-rise is acknowledged if the heel can be lifted at least 2 cm with stretched knee. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used 26.

   Ultrasound: The length between the calcaneus and the distal tip of the medial head of the gastrocnemius muscle.

   Amlangs ultrasound classification 27.

   Cost effectiveness analysis: A cost effectiveness analysis will be performed comparing the two treatment protocols.

   DVT screening: Ultra sound for deep Vein Thrombosis (DVT) will be performed after 2 and 8 weeks.

   Perimeter of calf: The perimeter of the calf is measured at the widest point on the injured side after 16 weeks. The distance from this point to lower edge of the patella is measured in centimeters. The distance is used to measure the perimeter on the healthy leg and for all subsequent measurements during the trial.

   Re-ruptur (RR): It is registered if the tendon re-ruptures during the trial period.

   Work: Hard physical labour involving heavy lifting, climbing stairs or climbing the ladder. E.g. bricklayer, paviour, carpenter, dustman, mailman.

   Moderate physical work that involves a lot of walking. E.g. salesperson, shop assistant, nurse.

   Light physical work which only involves light walking. E.g. office work

   Return to work: It is recorded how many days have passed before work is resumed part-time and full-time.

   Sport: Does the patient do sports? If yes, what kind, how many hours per week on average and at what level (professional, amateur, exerciser).

   Return to sport: It is recorded how many days have passed before sport activities are resumed and how many days have passed before sport activities reach a premorbid level.

   Health information: Former disease in or around the Achilles tendon, rheumatic disease, dominant leg.

   Other data: Age, Cpr.nr., other master data necessary to identify and call back the patient for post-examinations.

   The study is carried out in accordance with the principles of the Helsinki Declaration.

   Patients are covered by the patient insurance of Copenhagen University Hospital Hvidovre.

   The protocol as well as the patient information and declaration of consent must be approved by the National Committee on Health Research Ethics before inclusion of patients will begin.

   The project manager is responsible for informing the National Committee on Health Research Ethics of any critical adverse event and/or major changes of the protocol. All correspondence will be filed by the project manager.

   Declaration of consent All patients will receive verbal and written information concerning the study. The inclusion will take place after a declaration of consent has been obtained. It is the responsibility of the investigators to provide patients with comprehensive verbal and written information concerning the course of the study, purpose, potential risks and benefits.

   Statistics

   The two groups are described descriptively regarding demographic parameters as well as primary and secondary endpoints as described above in the paragraph "Data registration". Comparison of the primary and secondary outcomes of both groups is done by using relevant statistics according to the characteristics of the variables and if necessary the normal distribution. The change of the outcomes over a period of time is described within each group.

   The research group

   The study is carried out as collaboration between the research unit, Clinical Orthopaedic Research Hvidovre (www.corh.dk) and the Department of Physical- and Occupational Therapy, both at Copenhagen University Hospital Hvidovre.

   Data analysis and writing articles The data analysis and the drawing up of articles are done by the project manager and last-author. The project group is regularly involved in the process.

   Economic conditions

   The study is funded by the Department of Orthopaedic Surgery and the Department of Physiotherapy, Copenhagen University Hospital Hvidovre.

   The project group has independently initiated the study. Patients will not receive any fees for participation.

   Publication It is expected that the study will be published in an international, high-impact journal. We will furthermore seek to have the results presented at both national and international medical conventions. The results will also be published online and in other relevant media.

ELIGIBILITY:
Inclusion Criteria:

* rupture happened within 5 days.
* Age 18-70 years.
* The patient must be expected to be able to attend rehabilitation and post-examinations.
* The patient must be able to speak and understand Danish.
* The patient must be able to give informed consent.

Exclusion Criteria:

* Former rupture of one or both Achilles tendon(s).
* Previous surgery on the Achilles tendon.
* Fluoroquinolone treatment within the last 6 months.
* Tendinosis treated with corticosteroids (tablets or injections) within the last 6 months.
* The patient has been diagnosed with arterial insufficiency in the legs.
* Terminal illness or severe medical illness: ASA score higher than or equal to 3.
* The space between the rupture and the calcaneus is less than 1cm.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2014-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Achilles tendon Total Rupture Score | 12 months
  A patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture.

SECONDARY OUTCOMES:
Achilles tendon Total Rupture Score | 6 months
  A patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture.
Achilles tendon Total Rupture Score | 24 months
  A patient reported validation score developed to assess symptoms and physical activity after treatment for Achilles tendon rupture.
Heel-rise work test | 6 months
  Endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel-rises are counted and measured. The results are then compared to the weight of the patient and the total work is estimated. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used
Heel-rise work test | 12 months
  Endurance test where the patient stands on one leg and lifts the heel up and down until exhaustion. The number and the height of the heel-rises are counted and measured. The results are then compared to the weight of the patient and the total work is estimated. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used
Single heel-rise test | 6 months
  The patient stands with the foot in 10 degrees of dorsiflexion. It is recorded whether the patient is able to make a single heel-rise on the injured leg. The heel-rise is acknowledged if the heel can be lifted at least 2 cm with stretched knee. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used
Single heel-rise test | 12 months
  The patient stands with the foot in 10 degrees of dorsiflexion. It is recorded whether the patient is able to make a single heel-rise on the injured leg. The heel-rise is acknowledged if the heel can be lifted at least 2 cm with stretched knee. The MuscleLab ® (Ergo Test Technology, Oslo, Norway) measurement system is used
Ultrasound length measure | 6 months
  The length between the calcaneus and the distal tip of the medial head of the gastrocnemius muscle.
Ultrasound length measure | 12 months
  The length between the calcaneus and the distal tip of the medial head of the gastrocnemius muscle.
Cost effectiveness analysis | 12 months
  A cost effectiveness analysis will be performed comparing the two treatment protocols.
Re-rupture | 12 months
Re-rupture | 24 months
Perimeter of calf | 6 months
Perimeter of calf | 12 months
Return to work | 6 months
Return to work | 12 months
Return to work | 24 months
Return to sports | 6 months
Return to sports | 12 months
Return to sports | 24 months
Achilles Tendon Resting Angle (ATRA) | 6 months
Achilles Tendon Resting Angle (ATRA) | 12 months
Achilles Tendon Length Measure (ATLM) | 6 months
Achilles Tendon Length Measure (ATLM) | 12 months
Plantarflexion power | 6 months
  Plantarflexion power is measured with a hand held dynamometer fixed to the examination bed with a strong Velcro band.
Plantarflexion power | 12 months
  Plantarflexion power is measured with a hand held dynamometer fixed to the examination bed with a strong Velcro band.

OTHER OUTCOMES:
DVT screening | 2 and 8 weeks
  Ultra sound for deep Vein Thrombosis (DVT) will be performed after 2 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer W Barfod, MD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Copenhagen, Denmark

REFERENCES:
- [Derived] Barfod KW, Nielsen EG, Olsen BH, Vinicoff PG, Troelsen A, Holmich P. Risk of Deep Vein Thrombosis After Acute Achilles Tendon Rupture: A Secondary Analysis of a Randomized Controlled Trial Comparing Early Controlled Motion of the Ankle Versus Immobilization. Orthop J Sports Med. 2020 Apr 28;8(4):2325967120915909. doi: 10.1177/2325967120915909. eCollection 2020 Apr. PMID 32426409
- [Derived] Barfod KW, Hansen MS, Holmich P, Kristensen MT, Troelsen A. Efficacy of early controlled motion of the ankle compared with immobilisation in non-operative treatment of patients with an acute Achilles tendon rupture: an assessor-blinded, randomised controlled trial. Br J Sports Med. 2020 Jun;54(12):719-724. doi: 10.1136/bjsports-2019-100709. Epub 2019 Oct 9. PMID 31597624
- [Derived] Barfod KW, Hansen MS, Holmich P, Troelsen A, Kristensen MT. Efficacy of early controlled motion of the ankle compared with no motion after non-operative treatment of an acute Achilles tendon rupture: study protocol for a randomized controlled trial. Trials. 2016 Nov 29;17(1):564. doi: 10.1186/s13063-016-1697-2. PMID 27894329